CLINICAL TRIAL: NCT05482412
Title: Acute Paraphilic Pathway Down-Regulation In A Specialized Sensitive Group Using taVNS Modulation
Brief Title: Acute Intense Paraphilic Desire (DSM-V) Down-Regulation Via taVNS Neuro-Modulation [Transcutaneous Afferent Vagus Nerve] With Future Operative Implant Consideration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American University Of Montserrat (Other)
Collaborators: Greg Thomas William Consultant Research, Queens University (Unknown); Irene Becker Consultant, Coaching Certification for Pain Management (Unknown); Susan Jones MD PhD (Unknown); Peter Martin BSc Forensic Psych, Masters in Education, JPH Internal Meds + Family Meds Rotation Teaching Assistant (Unknown); Kofi McNair Nyamekye B Eng. Op. Neuromod. Masters + 4th Yr Meds Student (Unknown)
Responsible Party: Principal Investigator, Dr. Michel Rice, Associate Academic Dean Faculty of Medicine, Dean Research Department MD-PhD Program Faculty of Medicine, American University Of Montserrat
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHD1002
Record Dates: First submitted 2022-07-19; First posted 2022-08-01 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Desire; Sexual, Aversion; Paraphilia
Keywords: Down-Regulation; Vagus Cranial Nerve Modulation; Desire Control; taVNS [transcutaneous afferent vagus nerve stimulation]
MeSH Terms: conditions — Coitus; Paraphilic Disorders

STUDY DESIGN:
Intervention Model Description: The sequential study is involved in a translational study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Anonymity of participants is allowed for by using a participant computed platform assigning random visual stimulation sequences, thereby mixing Visual Inducer Test Media (T3, 4 & 5 (Young Adult)). The laboratory observer, software identification of participants, investigators, assessors & care providers are blinded in the software testing phase of the study.
  The taVNS intervention is also triple blinded (participant sham intervention, observer, care provider, investigators & assessors).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- T3 Subgroup (Experimental): Two T3 Subgroups:
  Paraphilia with androphilic or gynephilic Tanner 3 SI Marker (Sexual Incitation) note: incitation/stimulation
  Interventions: Device: transcutaneous (superficial) afferent electrical nerve stimulation specific for vagus nerve
- T5 (Young Adult) Subgroup (Experimental): Two T5 Subgroups Age-Play Subgroup (APSI):
  Paraphilia with androphilic or gynephilic Tanner 5 SI Marker (Sexual Incitation)
  Interventions: Device: transcutaneous (superficial) afferent electrical nerve stimulation specific for vagus nerve
- Sham Comparator (Sham Comparator): Medical Device Sham Comparator taVGN (Cranial Ten - Vagus Nerve) Selection of Random Participants In Any Subgroup Class Androphilic or gynephilic SI Marker (Sexual Incitation)
  Interventions: Device: transcutaneous (superficial) afferent electrical nerve stimulation specific for vagus nerve
- T2 Subgroup (Experimental): Two T2 Subgroups:
  Paraphilia with androphilic or gynephilic Tanner 2 SI Marker (Sexual Incitation)
  Interventions: Device: transcutaneous (superficial) afferent electrical nerve stimulation specific for vagus nerve
- T4 Subgroup (Experimental): Two T4 Subgroups:
  Paraphilia with androphilic or gynephilic Tanner 4 SI Marker (Sexual Incitation)
  Interventions: Device: transcutaneous (superficial) afferent electrical nerve stimulation specific for vagus nerve

INTERVENTIONS:
Device: transcutaneous (superficial) afferent electrical nerve stimulation specific for vagus nerve — Direct superficial auricular sensory branch of Cr X [Cranial Nerve Ten Vagus]

SUMMARY:
Transcutaneous Afferent Vagus Nerve Stimulation [taVNS] is used to modulate persistent & intense desire control amongst a specific participant group.

Testing Center Order of Deliver Number

DETAILED DESCRIPTION:
taVNS Diagnostic Spectrum Testing Center Order of Delivery

1. - Addiction - Opioid
2. - Chronic Pain - Central
3. - Anxiety + Panic Disorder
4. - MDD - Major Depression Disorder
5. - Addiction - Nicotine
6. - ADHD
7. - Addiction - Stimulant
8. - Addiction - Sexual + Love
9. - Addiction - Paraphilia
10. - Parkinsons
11. - Immune Enhancing
12. - Addiction - Overeating

RE-ORDERED CLINICAL TRIAL - NINE

Physiologic effects of taVNS stimulation have been extensively researched for over 150 years. Drug-resistant depression (MDD), migraine headaches, pelvic pain modulation, facilitation of motor learning in neonates, post stroke rehabilitation and seizures are some of the conditions investigated with favorable results using taVNS intervention. taVNS physiologic & mental effects have been noted to have advantageous therapeutic results on a vast diagnostic spectrum.

A clinical testing program for pre- and post-test was devised as a means to identify & measure treatment effects in specific T3, 4 and early 5 (Tanner) sub-group visual stimulation. The programmatic (software) of the stimulation medium created for this study is aimed to abate the use of a phallometric device purposed to measure sexual stimulation effects on participants.

Great effort has been assigned for the preservation of visual data to be shared in the investigators' research centre with other researchers internationally. The participant testing platform created for this study allows for a full-proof research ethics anonymous & confidential registry & testing process (triple blind).

Aggressive optimum (supra-threshold and below-pain threshold) taVNS is the therapeutic modality of choice in order to examine desire down-regulation effects using taVNS. DSM-V stock participants must be sub-grouped in the paraphilic categorical structure of the DSM-V.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 60 years old - heterosexual identifying as he/him

Exclusion Criteria:

* 35 to 40 age group - heterosexual identifying as he/him

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male identifying as he/him heterosexual
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual VITM Self-Reported Likert Scale for Desire (1 for no sexual inducement effect to 5 for intense sexual inducement effect) | Day 1 Intervention applied (atVNS) immediately after VITM testing if subject tested positive for desire in T4 subgroup
  Visual stimuli (VITM Visual Inducer Testing Media Software) used to measure desire (sexual fantasy) intensity as opposed to phallometric medium
Visual VITM Self-Reported Likert Scale for Desire (1 for no sexual inducement effect to 5 for intense sexual inducement effect)) | Day 1 Intervention applied (atVNS) immediately after VITM testing if subject tested positive for desire in T5 subgroup
  Visual stimuli (VITM Visual Inducer Testing Media Software) used to measure desire (sexual fantasy) intensity as opposed to phallometric medium
Visual VITM Self-Reported Likert Scale for Desire (1 for no sexual inducement effect to 5 for intense sexual inducement effect)) | Day 10 Intervention applied (atVNS) daily for 10 days followed by the VITM self-reported Likert Scale for Desire - T4 Subgroup
  Visual stimuli (VITM Visual Inducer Testing Media Software) used to measure desire (sexual fantasy) intensity as opposed to phallometric medium
Visual VITM Self-Reported Likert Scale for Desire (1 for no sexual inducement effect to 5 for intense sexual inducement effect)) | Day 10 Intervention applied (atVNS) daily for 10 days followed by the VITM self-reported Likert Scale for Desire - T5 Subgroup
  Visual stimuli (VITM Visual Inducer Testing Media Software) used to measure desire (sexual fantasy) intensity as opposed to phallometric medium

OTHER OUTCOMES:
Self-Reported Questionnaire | Day 1 Measured immediately post VITM testing of self-reported desire levels but before taVNS treatment
  Questions specific to participants' overall levels of desire intensity and distress in Likert Scale (1 no desire and 5 intense desire)
Self-Reported Questionnaire | Day 1 Measured immediately post VITM but post taVNS treatment
  Questions specific to participants' overall levels of desire intensity and distress in Likert Scale (1 no desire and 5 intense desire)
Self-Reported Questionnaire | Day 10 - After 10 treatments within 2 weeks) Measure immediately post VITM but post taVNS treatment
  Questions specific to participants' overall levels of desire intensity and distress in Likert Scale (1 no desire and 5 intense desire)

CONTACTS AND LOCATIONS:
Overall Officials: Athavan Gananathan, MD, Study Director — CEO AUM

IPD SHARING:
Plan to Share IPD: No
This study investigation began in 2015 during similar systematic review paper contractual work for international medical device manufacturers.
  This study involves sensitive subject matter requiring expected legal enforcements of research data collection and data/participant privacy protection.
  For these reasons, the data collected in this PhD study will not be shared.
  This research is owned by the University of Montserrat. VITM software is available for sharing without its sensitive materials for use by other researchers internationally. Please contact the University for more information.

REFERENCES:
- See also: Academy North Canada Division for American University of Montserrat — http://www.bettercalldoc.ca
- See also: Faculty of Medicine & University student information website — http://www.aummed.com